CLINICAL TRIAL: NCT03511898
Title: A Phase 1, Open-label, Multicenter, Dose Escalation Study to Evaluate the Safety of a Single Intravitreal Injection of THR-149 for the Treatment of Diabetic Macular Edema (DME)
Brief Title: A Study to Evaluate the Safety of THR-149 in Subjects With Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Organization: Oxurion (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: THR-149-001
Record Dates: First submitted 2018-04-10; First posted 2018-04-30 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- THR-149 dose level 1 (Experimental)
  Interventions: Drug: THR-149 dose level 1
- THR-149 dose level 2 (Experimental)
  Interventions: Drug: THR-149 dose level 2
- THR-149 dose level 3 (Experimental)
  Interventions: Drug: THR-149 dose level 3

INTERVENTIONS:
Drug: THR-149 dose level 1 — single intravitreal injection of THR-149 dose level 1
  Arms: THR-149 dose level 1
Drug: THR-149 dose level 2 — single intravitreal injection of THR-149 dose level 2
  Arms: THR-149 dose level 2
Drug: THR-149 dose level 3 — single intravitreal injection of THR-149 dose level 3
  Arms: THR-149 dose level 3

SUMMARY:
This study is conducted to evaluate the safety of a single intravitreal injection of THR-149.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Type 1 or type 2 Diabetes Mellitus
* Central-involved DME with central subfield thickness of ≥ 320µm on Spectralis® spectral domain optical coherence tomography (SD-OCT) or ≥ 305µm on non-Spectralis SD-OCT, in the study eye
* Best-corrected visual acuity (BCVA) ≤ 62 and ≥ 23 ETDRS letter score in the study eye
* Written informed consent obtained from the subject prior to screening procedures

Exclusion Criteria:

* Macular edema due to causes other than DME
* Concurrent disease in the study eye, other than central-involved DME, that could compromise BCVA, require medical or surgical intervention during the study period or could confound interpretation of the results
* Any condition that could confound the ability to detect a change in central subfield thickness in the study eye
* Previous confounding treatments / procedures, or their planned / expected use during the study period
* Presence of neovascularization at the disc (NVD) in the study eye
* Uncontrolled glaucoma in the study eye
* Any active ocular / intra-ocular infection or inflammation in either eye
* Poorly controlled Diabetes Mellitus
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities up to the Day 14 visit | up to Day 14

SECONDARY OUTCOMES:
Incidence of systemic and ocular adverse events including serious adverse events up to the end of the study | From Day 0 up to Day 84
Occurrence of laboratory abnormalities up to the end of the study | At Screening, Day 1, Day 7, Day 28 and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — ThromboGenics
Locations (7):
- United States (7):
  - Retina Consultants of Arizona, Phoenix, Arizona
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - Mid Atlantic Retina, Huntingdon Valley, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Retinal Research Center, PLLC, Austin, Texas
  - Retina Consultants of Houston, Houston, Texas